CLINICAL TRIAL: NCT06677047
Title: Assessment of Improvement in Functional Status of Patients With Pulmonary Fibrosis After Exercise Rehabilitation Program
Brief Title: Rehabilitation in Patients With Pulmonary Fibrosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Doctor, Assiut University
Other Study IDs: ILD& Rehabilitation
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the effects of exercise rehabilitation on the functional status of patients with pulmonary fibrosis, assessing both physical and psychological dimensions of health. By identifying significant improvements, we can contribute to the development of comprehensive rehabilitation strategies that enhance patient outcomes and foster a better quality of life for those affected by this challenging condition

DETAILED DESCRIPTION:
program is essential for understanding its efficacy. Functional status refers to an individual's ability to perform daily activities and maintain independence, which is particularly important for patients with chronic illnesses like PF. Evaluating changes in functional status not only helps in determining the success of rehabilitation efforts but also provides insights into the overall impact of exercise on patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1. **Diagnosis of Pulmonary Fibrosis:**
* Patients must have a confirmed diagnosis of pulmonary fibrosis, as determined by clinical evaluation and imaging studies (e.g., high-resolution computed tomography).

  2. **Age Range:**
* Participants should be adults aged 18 years and older to capture the adult population affected by the disease.

  3. **Stable Clinical Condition:**
* Patients must be in a stable clinical condition, defined as no exacerbations or significant changes in treatment for at least four weeks prior to enrollmen

Exclusion Criteria:

* 1. **Other Significant Lung Diseases:**
* Patients with concurrent respiratory conditions (e.g., chronic obstructive pulmonary disease, asthma, or lung cancer) that could confound the results.

  2. **Acute Exacerbations:**
* Individuals experiencing an acute exacerbation of pulmonary fibrosis or any significant respiratory illness within four weeks prior to enrollment.

  3. **Severe Comorbidities:**
* Patients with severe cardiovascular disease, uncontrolled hypertension, major neurological disorders, or musculoskeletal problems that would impede participation in exercise.

  4. **Cognitive Impairment:**
* Individuals with cognitive impairments that prevent them from understanding the study procedures or following the rehabilitation program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: **Demographic Data Collection:**
  * Age, sex, duration of pulmonary fibrosis, and medical history.
    2. **Pulmonary Function Testing:**
  * Spirometry will be conducted to assess Forced Vital Capacity (FVC) and Forced Expiratory Volume in one second (FEV1).
    3. **Functional Capacity Assessment:**
  * The Six-Minute Walk Test (6MWT) will be performed to evaluate baseline exercise tolerance.
    4. **Quality of Life Evaluation:**
  * Health-related quality of life will be assessed using the St. George's Respiratory Questionnaire (SGRQ) or Chronic Respiratory Disease Questionnaire (CRQ).
    5. **Dyspnea Assessment:**
  * Dyspnea levels will be measured using the Modified Medical Research Council (mMRC) dyspnea scale.
    * Exercise Rehabilitation Program
  Participants will engage in a structured 8-week exercise rehabilitation program, which includes:
  * **Supervised Exercise Sessions:**
  * Participants will attend twice-weekly sessions led by trained physiotherapists, focusing on aerobic
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
**Asses Health-Related Quality of Life:** | Baseline
  Assessed through validated questionnaires such as the St. George's Respiratory Questionnaire (SGRQ)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Troosters T, Janssens W, Demeyer H, Rabinovich RA. Pulmonary rehabilitation and physical interventions. Eur Respir Rev. 2023 Jun 7;32(168):220222. doi: 10.1183/16000617.0222-2022. Print 2023 Jun 30. PMID 37286219